CLINICAL TRIAL: NCT01553812
Title: The Assessment of Airway Resistance and Airtrapping in Elderly COPD Patients by Forced Oscillation Technique (FOT)
Status: Completed | Type: Observational
Sponsor: Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, Tse Hoi Nam, Resident Specialist, Kwong Wah Hospital
Other Study IDs: KW/EX-12-030 (48-15)
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: COPD
Keywords: forced oscillation technique; COPD; elderly; airway resistance; airtrapping
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The study hypothesize that parameters of new function machine---'forced oscillation technique' (FOT) can correlate well with the conventional lung function data for measurement of airway resistance and airtrapping in elderly COPD patients.

DETAILED DESCRIPTION:
INTRODUCTION:

Forced oscillation technique (FOT) may be a good supplementary tool to assess lung function in elderly since it is a simple and fast tool requiring minimal patients' cooperation.

AIMS:

To investigate the accuracy of forced oscillation test FOT in assessment of airway resistance and airtrapping in elderly COPD patients by comparing FOT parameters to various conventional lung function parameters including FEV1, FEF 25-75, RV/TLC ratio, IC etc. The best FOT parameter for airway resistance and airtrapping is also determined.

STUDY DESIGN:

A cross-sectional study conducted in Kwong Wah Hospital, Hong Kong, SAR

METHODS:

COPD patients were recruited from 1st Jan, 2010 to 31st Dec 2011. Both of the lung function tests (forced oscillation technique (FOT) and conventional lung function test) were performed. Parameters of FOT (FRes FDep, RAvr, XAvr, were compared with conventional lung function test for assessment of both airway resistance and airtrapping in COPD subjects. Adjusted FOT parameters (FResRatio and FDep) were also compared with %FEV1 and different GOLD stages.

Statistics:

Comparison between FOT parameters and spirometric parameters was done by correlation test and expressed as Spearman coefficient. ANOVA test is used to compare FOT parameters among different groups of GOLD stages (stage 1 to 4) and groups with various degree of airtrapping (stage 1 to 3). Post hoc analysis was estimated by Bonferroni test.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with previous lung function tests confirming irreversible obstructive pattern

Exclusion Criteria:

* Lung function test failed to show any obstructive pattern
* Paitents with co-existing pulmonary diseases including asthma, interstitial lung diseases, lung malignancy etc.
* Patients with active infectious diseases like tuberculosis

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients from both 'in-patient' and 'outpatient clinic' in Kwong Wah Hospital, Hong Kong, China
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

REFERENCES:
- [Derived] Tse HN, Tseng CZ, Wong KY, Yee KS, Ng LY. Accuracy of forced oscillation technique to assess lung function in geriatric COPD population. Int J Chron Obstruct Pulmon Dis. 2016 May 26;11:1105-18. doi: 10.2147/COPD.S102222. eCollection 2016. PMID 27307726